CLINICAL TRIAL: NCT00210574
Title: A Pilot Study of Topiramate in Childhood Absence Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR002872
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-04

CONDITIONS: Epilepsy, Absence
Keywords: childhood absence epilepsy; epilepsy; seizures; absence seizures
MeSH Terms: conditions — Epilepsy, Absence; Epilepsy; Seizures | interventions — Topiramate

INTERVENTIONS:
Drug: topiramate

SUMMARY:
Limited data exist on the effectiveness of antiepileptic drugs for treatment of childhood absence epilepsy. Preliminary data suggest that topiramate may be an effective drug for this condition. The present study is designed to provide further evidence of the potential effectiveness of topiramate for childhood absence epilepsy, as well as preliminary information about a potential target dose for future study.

DETAILED DESCRIPTION:
Childhood Absence Epilepsy (CAE) affects 2-11% of all children with epilepsy. CAE occurs most frequently in children between the ages of 4 and 10 years. Children with CAE have brief seizures (usually several seconds in duration) that typically involve staring and loss of awareness; twitching movement of the face or other areas of the body may also occur. Absence seizures are provoked by deep breathing for several minutes ("hyperventilation"). Topiramate is known to be effective in several types of seizures in children. Preliminary data from studies on other types of epilepsy, as well as case reports, suggest that it may also be effective in the type of seizures that occur in CAE. The objective of the study is to gather additional preliminary data on the effectiveness and the potential target dose of topiramate in CAE. Because CAE is not expected to resolve spontaneously in the age group being studied, no control group will be included. Patients in the study will receive increasing doses of topiramate, with the starting dose and dose increases at weekly intervals. The starting dose and dosage increases will be based on the child's weight. At each visit, hyperventilation will be used to determine if seizures can be provoked. If seizures occur, the dose will be further increased to the maximum dose for the study. If seizures do not occur with hyperventilation, an electroencephalogram (EEG) will be performed to confirm that the seizures are not occurring. If the EEG confirms that no seizures are occurring, topiramate dose will be maintained for 12 weeks. Topiramate will be given in the form of "sprinkles" contained within capsules that may be opened and the drug sprinkled onto food. Starting dose will depend on the child's weight, then increased to a maximum dose: 9 milligrams/kilogram/day or 400 milligrams/day, whichever is less for up to 162 days

ELIGIBILITY:
Inclusion Criteria:

* Weight of at least 15 kg (33 pounds)
* confirmed diagnosis of childhood absence epilepsy
* no other serious health problems or neurologic problems
* have not taken anti-epilepsy drugs other than ethosuximide, lamotrigine, or valproate
* able to take oral medication in a sprinkle capsule formulation
* girls must not have gotten their first menstrual period.

Exclusion Criteria:

* No seizures that are caused by something other than childhood absence epilepsy
* not taken topiramate, primidone, zonisamide, or phenobarbital in the past
* had to stop taking an anti-epilepsy drug (ethosuximide, lamotrigine, or valproate) because it was not effective in treating childhood absence epilepsy
* no presence of abnormal brain waves on electroencephalogram
* no presence of mental retardation, no autism, or severe developmental disorder.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2005-03; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who become seizure-free.

SECONDARY OUTCOMES:
Change in number of seizures per hour; change in duration of EEG spike wave discharges per hour; relationship between the lack of seizures and the blood level of topiramate.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A Pilot Study of Topiramate in Childhood Absence Epilepsy — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=497&filename=CR002872_CSR.pdf